CLINICAL TRIAL: NCT03993899
Title: Evaluation of the Impact of Coding the Fine Structure of the Sound on the Musical Perception in New Cochlear Implanted Subjects. Prospective Randomized Crossover Study.
Brief Title: Study of Quality Perception on Music in New Cochlear Implanted Subjects Using or Not a Fine Structure Strategy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: MED_EL_FS_music_Rennes_study
Record Dates: First submitted 2019-06-19; First posted 2019-06-21 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Sensorineural Hearing Loss, Bilateral
Keywords: cochlear implant stimulation strategy sound coding strategy
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Intervention Model Description: two arms A and B:
  Arm A: patient's fitting with strategy FS4 --> 15 days use --> tests and patient's fitting with strategy HDCIS --> 15 days use --> tests
  Arm B: patient's fitting with strategy HDCIS --> 15 days use --> tests and patient's fitting with strategy FS4 --> 15 days use --> tests
Who Masked: Participant, Investigator
Masking Description: Double blind study: the patient and the investigator don't know the strategy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cochlear implant (CI) with FineHearing Strategy then HDCIS (Active Comparator): cochlear implant with FineHearing strategy first during 15 days then with HDCIS strategy during 15 days
  Interventions: Device: FineHearing strategy or HDCIS strategy
- CI with HDCIS Strategy then FS4 (Active Comparator): cochlear implant with HDCIS strategy first during 15 days then with FS4 strategy during 15 days
  Interventions: Device: FineHearing strategy or HDCIS strategy

INTERVENTIONS:
Device: FineHearing strategy or HDCIS strategy — Cochlear implant with FineHearing strategy or HDCIS strategy

SUMMARY:
Main objective:

Show the superiority of Fine Structure (FS4) strategy compared to Continuous Interleaved Sampling (HDCIS) strategy on the qualitative preference for the listening of musical pieces.

Secondary objectives

* Show the superiority of FS4 strategy compared to the HDCIS strategy on the perception of musical elements (contour test).
* Analyze the link between the results of musical perception tests and the subjective preference of musical listening.
* Show the non inferiority of FS4 strategy compared to the HDCIS strategy on the perception of speech elements.
* Analyze the link between the results of musical perception tests and the results of the perception of speech elements.
* Analyze the qualitative multidimensional perception with HDCIS and FS4

DETAILED DESCRIPTION:
Introduction:

At present, most people with modern cochlear implant systems can understand speech using the device alone, at least under favorable listening conditions.

In recent years, research has increasing focussed on how implant users perceive sounds other than speech. In particular, music perception is of interest.

A review of the literature on musical perception with traditional implants, coding only the temporal envelope [McDermott 2004], revealed the following elements:

* On average, implant users perceive the rhythm approximately as well as listeners with normal hearing
* With technically sophisticated multi-channel sound processors, melody recognition, especially without rhythmic or verbal cues, is poor.
* The perception of timbre, especially the sounds of musical instruments, is generally unsatisfactory.
* Implant users tend to rate the quality of musical sounds as less enjoyable than listeners with normal hearing And studies show that the fine structure of sound is the main vector of information for music and the location of sounds. [Smith et al. 2002] It therefore seems necessary to focus on the contribution of the coding of the fine temporal structure of sound to the cochlear implant.

Main objective:

Show the superiority of FS4 strategy compared to HDCIS strategy on the qualitative preference for the listening of musical pieces.

Secondary objectives:

* Show the superiority of FS4 strategy compared to the HDCIS strategy on the perception of musical elements (contour test).
* Analyze the link between the results of musical perception tests and the subjective preference of musical listening.
* Show the non inferiority of FS4 strategy compared to the HDCIS strategy on the perception of speech elements.
* Analyze the link between the results of musical perception tests and the results of the perception of speech elements.
* Analyze the qualitative multidimensional perception with HDCIS and FS4

Plan of the study:

It is a prospective open monocentric randomized crossover study: measures will be done on the patient at 15 days and 30 days post-activation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥ 18 years old) speaking French
* Patient who fulfils the criteria for cochlear implantation

Exclusion Criteria:

- Retro-cochlear pathology: auditory neuropathy, vestibular schwannoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-01-07 (Actual)

PRIMARY OUTCOMES:
Qualitative measure of music | at 15 days post-activation
  The Gabrielsson scale (1988) is used to evaluate perceived sound quality as a multidimensional phenomenon, that is composed of a number of separate perceptual dimensions. Eight perceptual dimensions are evaluated: clarity, fullness, brightness vs dullness, hardness/sharpness vs softness, spaciousness, nearness, extraneous sounds, loudness. Visual analog scales (VAS) are used for each dimension and the patient has to score the dimension on a 10 cm VAS (between 0 to 10).
Qualitative measure of music | at 30 days post-activation
  The Gabrielsson scale (1988) is used to evaluate perceived sound quality as a multidimensional phenomenon, that is composed of a number of separate perceptual dimensions. Eight perceptual dimensions are evaluated: clarity, fullness, brightness vs dullness, hardness/sharpness vs softness, spaciousness, nearness, extraneous sounds, loudness. Visual analog scales are used for each dimension and the patient has to score the dimension on a 10 cm VAS (between 0 to 10).

SECONDARY OUTCOMES:
Speech recognition in quiet | at 15 days post-activation
  The speech recognition in quiet is evaluated with syllabic list of 40 phonemes. The patient has to recognize 21 syllables. The phonemes are scored: each good answer is scored 1 yielding a total between 0 and 1 (or 0% and 100%).
Speech recognition in quiet | at 30 days post-activation
  The speech recognition in quiet is evaluated with syllabic list of 40 phonemes. The patient has to recognize 21 syllables. The phonemes are scored: each good answer is scored 1 yielding a total between 0 and 1 (or 0% and 100%).
Differential frequency threshold | at 15 days post-activation
  This test aimed to determine the smallest perceptible difference in F0 between two stimuli for various baseline values of F0. An adaptive procedure is used.
Differential frequency threshold | at 30 days post-activation
  This test aimed to determine the smallest perceptible difference in F0 between two stimuli for various baseline values of F0. An adaptive procedure is used.
Melodic contour test | at 15 days post-activation
  The test stimuli of the melodic contour test (Galvin et al. 2007) are melodic contours composed of 5 notes of equal duration whose frequencies corresponded to musical intervals. Nine distinct musical patterns have to be identified by the patient. Each good answer is scored 1 yielding a total between 0 and 1 (or 0% and 100%).
Melodic contour test | at 30 days post-activation
  The test stimuli of the melodic contour test (Galvin et al. 2007) are melodic contours composed of 5 notes of equal duration whose frequencies corresponded to musical intervals. Nine distinct musical patterns have to be identified by the patient. Each good answer is scored 1 yielding a total between 0 and 1 (or 0% and 100%).

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Godey, Pr, Principal Investigator — Rennes University Hospital
Locations (1):
- CHU Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No